CLINICAL TRIAL: NCT04964947
Title: Does Prophylactic Local Tobramycin Injection Lower Open Fracture Infection Rates?
Brief Title: Tobramycin Injection to Prevent Infection in Open Fractures
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arun Aneja, MD, PhD, Orthopaedic Trauma Surgeon, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P003263; GRANT13200494 (Other Grant/Funding Number: DOD, Department of Defense)
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Wound Infection; Fractures, Open; Surgical Site Infection
Keywords: Local antibiotic; Non-union; Aminoglycoside; Tobramycin; Open extremity fracture; fracture related infection
MeSH Terms: conditions — Wound Infection; Fractures, Open; Surgical Wound Infection | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tobramycin Treatment Group (Experimental): Participants in this group receive a local aqueous tobramycin injection (2mg/mL) plus standard of care treatment.
  Interventions: Drug: Tobramycin Injection
- Standard of Care Treatment Group (No Intervention): Participants in this group receive standard of care treatment.

INTERVENTIONS:
Drug: Tobramycin Injection — 80 milligrams of tobramycin diluted in 40 milliliters of normal saline
  Arms: Tobramycin Treatment Group

SUMMARY:
The goal of open extremity fracture (OEF) treatment is to promote fracture healing and restore function while preventing the development of infection. This is achieved through systematic and timely wound debridement and irrigation, fracture stabilization, tetanus prophylaxis, systemic and local antimicrobial therapy, and judicious timing of wound closure based on cleanliness. Early prophylactic systemic antibiotics lower infection rates in open fractures but have limitations of achieving adequate concentration at the hypoperfused wound area. OEF wounds are frequently poor in vasculature secondary to the soft tissue injury, hence adequate concentration of antibiotic cannot permeate to the tissue at risk. If systemic antibiotic concentrations are increased to achieve minimum inhibitory concentration (MIC) for pathogens at the wound, there is heightened concern for systemic drug toxicity. In sharp contrast, locally administered antibiotics achieve high drug concentration directly within the wound cavity with minimal systemic side effects. Local antibiotic therapy has shown to reduce rates of open fracture wound infection. With the serious implications of postoperative infections in OEF, it is imperative that all measures including further use of prophylactic local antibiotics be considered to prevent fracture-related infection (FRI). The overarching hypothesis for this project is that a novel synergistic combination of local aqueous tobramycin plus perioperative weight-based IV cephalosporin antibiotic prophylaxis will reduce the rate of FRI one year after OEF surgery. This in turn will improve OEF patient outcomes, decreasing morbidity and return to the operating room (OR) without any adverse effect on fracture healing. Regardless of the treatment group, bacterial speciation will be determined for patients that do develop FRI to help guide future treatment. The goal is to improve the clinical outcome and recovery of the population that sustains an OEF by decreasing the rate of FRI and fracture nonunions while concurrently educating on bacterial speciation and resistance.

ELIGIBILITY:
Inclusion Criteria:

* Open fracture to arm, leg, or both
* Over the age of 18

Exclusion Criteria:

* Under the age of 18
* Allergy to tobramycin or any other antibiotic in the aminoglycoside family
* Previously treated with a resorbable antibiotic carrier
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rate of infection | 1 year
  Rate of infection one year after open fracture fixation surgery.

SECONDARY OUTCOMES:
Tobramycin effects on non-union | 3 months after surgery
  Modified radiographic union score for tibial fracture (mRUST) scores combined with clinical observation of functional weight bearing at 3 months will be assessed. If union status remains unclear, nonunion will be further defined as a need for secondary bone grafting or surgical intervention.
Tobramycin effects on non-union | 6 months after surgery
  Modified radiographic union score for tibial fracture (mRUST) scores combined with clinical observation of functional weight bearing at 6 months will be assessed. If union status remains unclear, nonunion will be further defined as a need for secondary bone grafting or surgical intervention.
Tobramycin effects on non-union | 12 months after surgery
  Modified radiographic union score for tibial fracture (mRUST) scores combined with clinical observation of functional weight bearing at 12 months will be assessed. If union status remains unclear, nonunion will be further defined as a need for secondary bone grafting or surgical intervention.
Difference in bacterial specification between treatment and standard of care group. | 12 months
  Upon identification of a fracture-related infection within the first 12 months following surgical fixation, sterile intraoperative cultures will be obtained and grown over 21 days to determine bacterial speciation.
Difference in antibiotic resistance between treatment and standard of care group. | 12 months
  Upon identification of a fracture-related infection within the first 12 months following surgical fixation, sterile intraoperative cultures will be obtained and grown over 21 days to determine antimicrobial resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Aneja, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pilot Study Results — https://journals.lww.com/jorthotrauma/abstract/9900/does_local_aqueous_tobramycin_injection_reduce.388.aspx